CLINICAL TRIAL: NCT02390921
Title: The Effectiveness of Oral Treatment With Liposomated Iron in Patients With Previous Bariatric Surgery Which Are Currently Receiving Chronic Parentheral Therapy With Iron
Brief Title: The Use of Liposomated Iron After Bariatric Surgery in Patients That Are Receiving Parentheral Therapy With Iron
Acronym: BARIFER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR(AG)275/2014
Record Dates: First submitted 2015-02-05; First posted 2015-03-18 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Liposomated Iron; Y-de-Roux Gastric By-Pass; Parenteral Iron Therapy
MeSH Terms: interventions — Therapeutics; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liosomated iron therapy (Active Comparator): Fisiogen Ferro Forte 28mg every day po, during 3 months
  Interventions: Drug: Fisiogen Ferro Forte
- Endovenous Iron Therapy (Experimental): Venofer 300mg endovenously every 3 months
  Interventions: Drug: Venofer

INTERVENTIONS:
Drug: Fisiogen Ferro Forte — The patients will interrupt the endovenous treatment with iron and will receive liposomated iron 28mg/daily during 3 months.
  Other Names: Oral treatment with liposomated iron (Fisiogen Ferro Forte)
  Arms: Liosomated iron therapy
Drug: Venofer — The patients will continue their usual endovenous administration of Venofer 300mg every 3 month
  Other Names: Endovenous treatment with Venofer 300mg every 3 month
  Arms: Endovenous Iron Therapy

SUMMARY:
Bariatric surgery is the most effective long-term treatment of morbid obesity treatment, so you can maintain weight loss enduringly with improvement or resolution of comorbidity and mortality reduction. All bariatric surgery techniques in postoperative induce a significant reduction in food intake and / or absorption of nutrients and therefore may be associated with a risk of nutritional deficiency, which increases over the years after surgery. One of the nutrients whose absorption is affected significantly is iron, women of childbearing age segment most vulnerable being. A significant percentage of these women require oral supplementation with high doses of iron and often parenteral treatment is needed for digestive intolerance or therapeutic failure.

Hypothesis: The liposome orally administered iron could represent a therapeutic alternative in women of childbearing age, previously undergone bariatric surgery that currently require parenteral iron therapy.

Objectives: To evaluate the tolerability and efficacy of oral iron liposome female patients previously undergone bariatric surgery that currently require parenteral replacement therapy, as well as the impact on quality of life.

Methods: a single center, open, prospective, interventional, in 40 women of childbearing age, previously undergone bariatric surgery, which currently require intravenous iron therapy chronically. Subjects will be divided into 2 parallel groups: 20 cases and 20 controls matched for age, level of Hb, year after surgery and percentage of weight lost.

Relevance: This study will allow us to identify an alternative treatment with oral iron in the case of patients with severe iron deficiency after bariatric surgery, which currently require parenteral iron therapy due to intolerance to current oral products or therapeutic failure. At the same time it could help reduce healthcare costs and improve the quality of life of these patients, who will not have to enter periodically in solitary day hospital for administration of parenteral iron.

DETAILED DESCRIPTION:
This project is proposed with the aim of exploring the efficacy and tolerability of liposome orally administered iron in female patients previously undergone bariatric surgery (gastric bypass) currently receiving parenteral iron therapy chronically.

The hypotheses are:

(i) .- A significant percentage of patients undergoing bariatric surgery have iron deficiency and chronic complication. In the investigators series, approximately 100 women require intravenous iron therapy in a chronic (10% of all patients undergoing bariatric surgery to date), significantly increasing costs.

(ii) .- The liposomal form of iron does not depend on gastric pH and increased bioavailability is not dependent on the presence of the digestive dudodeno circuit.

(iii) .- Increased iron absorption and tolerability allow us to remove chronic intravenous iron therapy in the case of these patients. Thus, majoraria quality of life by reducing healthcare costs and avoiding adverse reactions associated with the procedure.

Main objective: To evaluate the tolerability and efficacy of oral iron liposome female patients previously undergone bariatric surgery that currently require parenteral replacement therapy for chronic form.

Secondary objectives:

(i) .- To evaluate the change in the levels of Hb, ferritin, iron, transferrin saturation at 4, 12 weeks of treatment.

(ii) .- Lay the foundation for future study of pharmacokinetics and pharmacodynamics in patients undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* In the clinical study will include:

  * women who underwent Y-de-Roux gastric by-pass
  * over 18 years, premenopausal
  * stable weight in the previous 6 months
  * currently receiving parenteral iron therapy regularly in solitary day hospital
  * which have signed the informed consent

Exclusion Criteria:

* male
* with mobility problems that constrain a marked inactivity
* with associated disease (chronic obstructive pulmonary cardiac cerebral vascular-disease, illness, accident sequel , severe psychiatric or eating disorder
* undergoing different surgical techniques to gastric bypass
* other causes of iron deficiency.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Non-inferiority (change in the levels of Hemoglobin) | 3 months
  To evaluate the change in the levels of Hemoglobin at 4 and 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andreea Ciudin, Principal Investigator — Vall d´Hebron University Hospital
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No